CLINICAL TRIAL: NCT06827587
Title: Efficacy, Safety, and PKPD Study of Efgartigimod Sequential Therapy with Telitacicept in Generalized Myasthenia Gravis (gMG): an Open-label, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Efgartigimod Sequential Therapy with Telitacicept in Generalized Myasthenia Gravis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-298
Record Dates: First submitted 2025-01-23; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Myasthenia Gravis; Autoimmune Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases; Neuromuscular Diseases | interventions — telitacicept; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Efgartigimod + Telitacicept (1-week interval) group (Experimental): Starting from Week 0, participants will receive efgartigimod (10 mg/kg) for induction treatment by intravenous infusion over 1 hour, administered once a week for 4 consecutive weeks.
  After a 1-week interval, at Week 5, participants will receive telitacicept (240 mg) for maintenance treatment, administered once a week by subcutaneous injection for a total of 25 weeks.
  Follow-up will continue until Week 30.
  Interventions: Drug: Efgartigimod + Telitacicept (1-week interval) group
- Efgartigimod + Telitacicept (2-week interval) group (Experimental): Starting from Week 0, participants will receive efgartigimod (10 mg/kg) for induction treatment by intravenous infusion over 1 hour, administered once a week for 4 consecutive weeks.
  After a 2-week interval, at Week 6, participants will receive telitacicept (240 mg) for maintenance treatment, administered once a week by subcutaneous injection for a total of 24 weeks.
  Follow-up will continue until Week 30.
  Interventions: Drug: Efgartigimod + Telitacicept (2-week interval) group
- Telitacicept-only group (Active Comparator): Participants will not receive efgartigimod for induction treatment. Starting from Week 0, participants will receive telitacicept (240 mg) for maintenance treatment, administered once a week by subcutaneous injection for a total of 30 weeks.
  Follow-up will continue until Week 30.
  Interventions: Drug: Telitacicept-only group

INTERVENTIONS:
Drug: Efgartigimod + Telitacicept (1-week interval) group — Drug 1: Efgartigimod
  Generic Name: Efgartigimod Formulation: Injection (Intravenous) Dose: 10 mg/kg Frequency: Once a week Route of Administration: Intravenous infusion Duration: 4 weeks (Week 0 to Week 4) Drug 2: Telitacicept
  Generic Name: Telitacicept Formulation: Injection (Subcutaneous) Dose: 240 mg Frequency: Once a week Route of Administration: Subcutaneous injection Duration: 25 weeks (Week 5 to Week 29)
  Other Names: E+1w+T
  Arms: Efgartigimod + Telitacicept (1-week interval) group
Drug: Efgartigimod + Telitacicept (2-week interval) group — Drug 1: Efgartigimod
  Generic Name: Efgartigimod Formulation: Injection (Intravenous) Dose: 10 mg/kg Frequency: Once a week Route of Administration: Intravenous infusion Duration: 4 weeks (Week 0 to Week 4) Drug 2: Telitacicept
  Generic Name: Telitacicept Formulation: Injection (Subcutaneous) Dose: 240 mg Frequency: Once a week Route of Administration: Subcutaneous injection Duration: 24 weeks (Week 6 to Week 29)
  Other Names: E+2w+T
  Arms: Efgartigimod + Telitacicept (2-week interval) group
Drug: Telitacicept-only group — Drug: Telitacicept Generic Name: Telitacicept Formulation: Injection (Subcutaneous) Dose: 240 mg Frequency: Once a week Route of Administration: Subcutaneous injection Duration: 30 weeks (Week 0 to Week 29)
  Other Names: T-only
  Arms: Telitacicept-only group

SUMMARY:
Title: The Efficacy, Safety, and PK/PD of Efgartigimod Followed by Telitacicept in Generalized Myasthenia Gravis: Protocol of a Randomized Controlled Trial Objective: This study aims to evaluate the efficacy, safety, and pharmacokinetics/pharmacodynamics (PK/PD) of efgartigimod followed by telitacicept in patients with generalized myasthenia gravis (gMG). Specifically, the trial seeks to determine the optimal treatment strategy for gMG by assessing the effect of sequential biologic therapy on disease management.

Study Design: This is a multi-center, open-label, randomized controlled trial involving 60 acetylcholine receptor antibody-positive gMG patients.

DETAILED DESCRIPTION:
Study Overview: This study is a multi-center, open-label, randomized controlled trial designed to evaluate the efficacy, safety, and pharmacokinetics/pharmacodynamics (PK/PD) of a sequential treatment regimen combining efgartigimod followed by telitacicept in patients with generalized myasthenia gravis (gMG). The trial aims to determine whether the sequential use of these two biologics provides enhanced therapeutic benefits compared to monotherapy and to identify the optimal interval between treatments.

Background: Generalized myasthenia gravis (gMG) is an autoimmune neuromuscular disorder primarily characterized by skeletal muscle weakness and fatigue due to pathogenic autoantibodies, most commonly against acetylcholine receptors (AChR). While conventional treatments for gMG include cholinesterase inhibitors, steroids, and immunosuppressants, biologic therapies have shown great promise in addressing the underlying autoimmune mechanisms.

New biologics, such as efgartigimod (a neonatal Fc receptor inhibitor) and telitacicept (a BLyS/APRIL inhibitor), have demonstrated efficacy in treating gMG, but the optimal sequencing and duration of their use have not been thoroughly explored. Efgartigimod, which accelerates the depletion of pathogenic IgG antibodies, has shown quick symptom relief but with a relatively short duration of effect. Telitacicept, an antibody fusion protein that inhibits BLyS and APRIL to suppress B-cell maturation, has demonstrated potential for longer-term disease control. This trial seeks to evaluate the sequential combination of these two biologics, specifically exploring the best interval between treatments.

Study Design: This study is designed to explore the efficacy, safety, and PK/PD characteristics of efgartigimod followed by telitacicept in patients with AChR-Ab-positive generalized myasthenia gravis (gMG). The trial will enroll 60 patients who are randomized into three groups:

Efgartigimod + Telitacicept (1-week interval) group (E+1w+T) Efgartigimod + Telitacicept (2-week interval) group (E+2w+T) Telitacicept-only group (T only) The trial will be conducted at five clinical centers, with a study period from February 2025 to February 2026.

Treatment Regimens:

Efgartigimod + Telitacicept Sequential Therapy:

Efgartigimod (10 mg/kg) will be administered intravenously once per week for 4 weeks. Following a 1-week or 2-week break after the efgartigimod treatment, telitacicept (240 mg) will be administered subcutaneously once per week for a total of 24-25 weeks.

Telitacicept-only Group:

Patients in the Telitacicept-only group (T only) will receive telitacicept (240 mg) subcutaneously once a week for 30 weeks, without prior treatment with efgartigimod.

Primary and Secondary Endpoints:

Primary Endpoint: The primary endpoint of this study is the change from baseline in the Quantitative Myasthenia Gravis (QMG) score at Week 30. The QMG score is a validated clinical measure used to assess the severity of myasthenia gravis symptoms.

Secondary Endpoints:

Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) score.

The proportion of patients achieving minimal manifestation status (MMS) is defined as having no significant functional impairment despite observable weakness.

Change in steroid and immunosuppressant doses at Weeks 24 and 30. Incidence of MG exacerbations, myasthenic crises, and adverse events. PK/PD characteristics of telitacicept, including blood drug concentration, B-cell counts, and levels of BLyS/APRIL.

Pharmacokinetics and Pharmacodynamics:

Pharmacokinetics (PK) includes testing the blood concentration, clearance（CI）, and distribution volume of telitacicept, and pharmacodynamics (PD) includes testing serum immunoglobulins, B cell counts, and/or Blys+APRIL levels.

IgG levels will be assessed at baseline, after 4 weeks of efgartigimod treatment, and during telitacicept therapy to monitor the drug's pharmacodynamic effects on immune parameters.

Safety Monitoring:

Safety will be assessed by recording the incidence of adverse events (AEs), serious adverse events (SAEs), and any other clinically relevant changes in laboratory values or vital signs.

NCI-CTCAE v5.0 will be used to grade the severity of adverse events. Telitacicept will be administered cautiously, with specific attention to potential infections or autoimmune complications, given its mechanism of action on B cells.

Exploratory and Additional Analyses:

An exploratory analysis will evaluate whether the sequencing and timing of efgartigimod and telitacicept impacts the long-term disease control in gMG patients.

The study will also assess how the sequential administration of efgartigimod and telitacicept compares to telitacicept-only therapy in terms of symptom control and reduction in disease-related markers.

Statistical Methods:

The study uses Analysis of Covariance (ANCOVA) to compare changes from baseline in QMG scores between the treatment groups.

The statistical analysis will follow the Intention-to-treat (ITT) principle, with efficacy measured in the Full Analysis Set (FAS) and safety in the Safety Analysis Set (SS).

Sample Size: Each treatment group is expected to enroll 20 patients, accounting for a 15% dropout rate, bringing the total sample size to 60 patients (20:20:20).

Power Analysis: The study is powered at 80% to detect a 4-point improvement in QMG score between the sequential treatment groups and the Telitacicept-only group, with a significance level of α=0.025.

Discussion:

This study is the first to explore sequential biologic therapy using efgartigimod followed by telitacicept in generalized myasthenia gravis.

The study builds on prior research showing the efficacy and safety of both drugs individually, but it is the first to explore their combined use in a sequential regimen.

Given that efgartigimod and telitacicept have different mechanisms of action-efgartigimod rapidly depleting IgG autoantibodies and telitacicept inhibiting B-cell maturation-the combination is expected to offer long-term symptom relief, with the potential to reduce the need for other immunosuppressive therapies.

This trial will help determine the optimal timing for sequential administration, providing important insights for future treatment strategies in gMG patients.

Study Limitations:

As this is a pilot exploratory trial, the results should be interpreted cautiously due to the relatively small sample size.

Follow-up will be limited to 30 weeks, which may not capture the full long-term effects and safety profile of the combination therapy.

Conclusion:

The efgartigimod followed by telitacicept sequential therapy has the potential to significantly improve the treatment of gMG, offering a new approach to managing patients who have previously experienced inadequate symptom control with conventional therapies. The results from this study could provide crucial evidence for the development of a robust sequential biologic treatment strategy for gMG.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily signs the informed consent form.
* Age ≥18 and ≤80 years, regardless of gender.
* Meets the diagnostic criteria for Myasthenia Gravis (MG) as per the 2020 China MG Diagnosis and Treatment Guidelines, with serological evidence of positive AChR-Ab.
* MG Clinical Classification according to the Myasthenia Gravis Foundation of America (MGFA) Staging System: Grade II-IV.
* Patients with fluctuating MG symptoms before enrollment, as indicated by MG-ADL score ≥6 or Quantitative Myasthenia Gravis score (QMG) ≥8, maintained for more than 24 hours.

Exclusion Criteria:

* Coexisting active autoimmune diseases, such as Systemic Lupus Erythematosus (SLE), Rheumatoid Arthritis, Sjögren's Syndrome, etc.
* Patients with active infections, such as Herpes Zoster, HIV, active Tuberculosis, active Hepatitis.
* Patients with thymoma who have undergone surgery within the past 6 months.
* Patients with malignancies other than thymoma.
* Patients with severe liver or renal dysfunction, defined as: Liver function: ALT or AST > 3 ×ULN (upper limit of normal). Renal function: Glomerular filtration rate (GFR) < 30 mL/min/1.73m².
* IgG ≤ 400 mg/dL.
* Patients who have used biologic agents before enrollment and are within 5 half-lives of the drug, such as those who have used Telitacicept within the past 2 months, Efgartigimod within the past 1 month, or Rituximab within the past 6 months.
* Patients who have received intravenous immunoglobulin (IVIg) or undergone plasmapheresis within the past 2 months before enrollment.
* Patients who have received any live vaccines within 3 months before the study or plan to receive any vaccines during the study.
* Pregnant or breastfeeding women, or those planning to conceive during the trial.
* Patients with allergies to human-derived biologics.
* Patients who have participated in any clinical trial within the 28 days before enrollment or are within 5 half-lives of the investigational drug used in a prior clinical trial.
* Other patients deemed unsuitable for enrollment by the investigator (e.g., severe mental disorders).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in QMG score | 30 weeks after randomization
  Change in QMG score from baseline to Weeks 30. Total QMG scores range from 0 (none) to 39 (severe).

SECONDARY OUTCOMES:
Change from baseline in MG-ADL score | Weeks 4, 8, 12, 18, 24, and 30 after randomization.
  Change in Myasthenia Gravis Activities of Daily Living (MG-ADL) score from baseline at weeks 4, 8, 12, 18, 24, and 30. Total MG -ADL scores range from 0 (normal) to 24 (severe).
Proportion of subjects with minimal manifestation status (MMS) | 4, 8, 12, 18, 24, and 30 weeks after randomization.
  Proportion of patients achieving minimal status (MMS) at weeks 4, 8, 12, 18, 24, and 30 (MMS is defined as the absence of any functional limitations due to myasthenia, although mild myasthenia may be detected upon examination by a specialized neuromuscular physician).
Proportion of subjects with a ≥2-point reduction in MG-ADL score from baseline | 4, 8, 12, 18, 24, and 30 weeks after randomization.
  Proportion of subjects in each group with a decrease of ≥2 points in MG-ADL .score from baseline at weeks 4, 8, 12, 18, 24, and 30.
Proportion of subjects with a ≥3-point reduction in QMG score from baseline | 4, 8, 12, 18, 24, and 30 weeks after randomization.
  Proportion of subjects in each group with a decrease of ≥3 points in QMG score from baseline at weeks 4, 8, 12, 18, 24, and 30.
Changes in the doses of steroids and other immunosuppressants | 24 and 30 weeks after randomization.
  Changes in the doses of steroids and other immunosuppressants from baseline at weeks 24 and 30
Proportion of patients with a prednisone (or equivalent corticosteroid) dose ≤5 mg/day | 24 and 30 weeks after randomization.
  Proportion of patients with a prednisone (or equivalent corticosteroid) dose ≤5 mg/day at weeks 24 and 30.
Incidence of MG relapse/acute exacerbation and myasthenic crisis | Week 30 after randomization
  Incidence of MG relapse/acute exacerbation and myasthenic crisis at week 30
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Week 30 after randomization
  Incidence of adverse events (AEs) and serious adverse events (SAEs) at week 30. The assessment of adverse events will be conducted according to the Common Terminology Criteria for Adverse Events (CTCAE) V5.0, as defined by the National Cancer Institute (NCI).

OTHER OUTCOMES:
Plasma concentration of telitacicept in the two sequential treatment groups | 30 minutes before the first dose of telitacicept, and 6 hours, 24 hours, 48 hours, 72 hours, Week 1, Week 4, Week 8, Week 12, and Week 24 after the first dose.
  The study will measure the plasma concentration of telitacicept in patients receiving the sequential treatment regimen. Blood samples will be collected at the following time points: 30 minutes before the first dose, 6 hours ± 15 minutes post-dose, 24 hours ± 1 hour (1 day), 48 hours ± 2 hours (2 days), 72 hours ± 3 hours (3 days), pre-dose at Week 1 ± 12 hours, pre-dose at Week 4 ± 3 days, and pre-dose at Week 8 ± 3 days. Subsequently, blood samples will be collected every 3 months before each telitacicept dose at the following time points: pre-dose at Week 12 ± 3 days and pre-dose at Week 24 ± 3 days.
Serum immunoglobulins | At baseline, after one cycle (4 weeks) of efgartigimod treatment, before the first dose of telitacicept, and at Week 1, Week 4, and every subsequent 4-week interval after the first dose of telitacicept
  Serum immunoglobulin levels, as a pharmacodynamic marker for both efgartigimod and telitacicept, will be measured at baseline, after 1 cycle (4 weeks) of efgartigimod treatment, before the first dose of telitacicept, and at Weeks 1, 4, and every subsequent 4-week interval after telitacicept administration.
B-cell subpopulation count and BLyS/APRIL measurement | Before the first dose of telitacicept, at Week 4, at Week 12, and at Week 24.
  B-cell subpopulation count and BLyS/APRIL measurement will be performed before the first dose of telitacicept and before dosing at Week 4, Week 12, and Week 24.
Clearance(CI) of telitacicept in the two sequential treatment groups | 30 minutes before the first dose of telitacicept, and 6 hours, 24 hours, 48 hours, 72 hours, Week 1, Week 4, Week 8, Week 12, and Week 24 after the first dose.
  The study will measure the clearance(CI) of telitacicept in patients receiving the sequential treatment regimen. Blood samples will be collected at the following time points: 30 minutes before the first dose, 6 hours ± 15 minutes post-dose, 24 hours ± 1 hour (1 day), 48 hours ± 2 hours (2 days), 72 hours ± 3 hours (3 days), pre-dose at Week 1 ± 12 hours, pre-dose at Week 4 ± 3 days, and pre-dose at Week 8 ± 3 days. Subsequently, blood samples will be collected every 3 months before each telitacicept dose at the following time points: pre-dose at Week 12 ± 3 days and pre-dose at Week 24 ± 3 days.
Volume of distribution (Vd) of telitacicept in the two sequential treatment groups | 30 minutes before the first dose of telitacicept, and 6 hours, 24 hours, 48 hours, 72 hours, Week 1, Week 4, Week 8, Week 12, and Week 24 after the first dose.
  The study will measure the volume of distribution (Vd) of telitacicept patients receiving the sequential treatment regimen. Blood samples will be collected at the following time points: 30 minutes before the first dose, 6 hours ± 15 minutes post-dose, 24 hours ± 1 hour (1 day), 48 hours ± 2 hours (2 days), 72 hours ± 3 hours (3 days), pre-dose at Week 1 ± 12 hours, pre-dose at Week 4 ± 3 days, and pre-dose at Week 8 ± 3 days. Subsequently, blood samples will be collected every 3 months before each telitacicept dose at the following time points: pre-dose at Week 12 ± 3 days and pre-dose at Week 24 ± 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, Bachelor, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Zhang Y, Deng Y, Li W, Wang Y, Qi F, Zhang Q, Wan B, Li X, Weng Y, Fang Z, Zhang Y, Qu X, Pan S, Yang S, Zhang X. The efficacy, safety, and pharmacokinetics/pharmacodynamics of telitacicept following efgartigimod in generalized myasthenia gravis: protocol of a randomized controlled trial. Front Immunol. 2025 Oct 22;16:1604786. doi: 10.3389/fimmu.2025.1604786. eCollection 2025. PMID 41200184